CLINICAL TRIAL: NCT02382848
Title: Effectiveness of Prazosin in Bulimic Patients Experiencing Nightmares Due to PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Fauzia Mahr, MD, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00001746
Record Dates: First submitted 2015-02-18; First posted 2015-03-09 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Stress Disorders, Post-Traumatic; Bulimia Nervosa
Keywords: Eating Disorders; Bulimia Nervosa; Nightmares; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Bulimia Nervosa; Feeding and Eating Disorders | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prazosin, Then Placebo (Active Comparator): Participants first received Prazosin. A starting dose of Prazosin (1mg capsule) will be given at Week # 1 of this arm. Symptoms will be reassessed and medication will be adjusted by 1-2 mg increments every 7 days for 3 weeks based on clinical response and severity of night mares, to achieve maximum therapeutic benefit while monitoring adverse effects using side effects scale on weekly basis (psychiatrist will be using the scale at every visit). The end point for capping the Prazosin dose will be 6 mg daily. After a washout period, they then receive Placebo
  Interventions: Drug: Prazosin; Drug: Placebo
- Placebo, Then Prazosin (Placebo Comparator): Participants first received Placebo (matching Prazosin) for a 3 consecutive week period during the 7 week study period. After a washout period, they then received Prazosin. The starting dose of Prazosin (1mg capsule) will be given at Week # 5 of this arm. Symptoms will be reassessed and medication will be adjusted by 1-2 mg increments every 7 days for 3 weeks based on clinical response and severity of night mares, to achieve maximum therapeutic benefit while monitoring adverse effects using side effects scale on weekly basis (psychiatrist will be using the scale at every visit). The end point for capping the Prazosin dose will be 6 mg daily.
  Interventions: Drug: Prazosin; Drug: Placebo

INTERVENTIONS:
Drug: Prazosin — A starting dose of Prazosin (1mg capsule) will be given at Week # 1 of this arm. Symptoms will be reassessed and medication will be adjusted by 1-2 mg increments every 7 days for 3 weeks based on clinical response and severity of night mares, to achieve maximum therapeutic benefit while monitoring adverse effects using side effects scale on weekly basis (psychiatrist will be using the scale at every visit). The end point for capping the Prazosin dose will be 6 mg daily.
  Arms: Prazosin, Then Placebo
Drug: Placebo — Prazosin-matched placebo pill
  Arms: Prazosin, Then Placebo
Drug: Prazosin — A starting dose of Prazosin (1mg capsule) will be given at Week # 5 of this arm. Symptoms will be reassessed and medication will be adjusted by 1-2 mg increments every 7 days for 3 weeks based on clinical response and severity of night mares, to achieve maximum therapeutic benefit while monitoring adverse effects using side effects scale on weekly basis (psychiatrist will be using the scale at every visit). The end point for capping the Prazosin dose will be 6 mg daily.
  Arms: Placebo, Then Prazosin
Drug: Placebo — Prazosin-matched placebo pill
  Arms: Placebo, Then Prazosin

SUMMARY:
This research is being done to find out how effective Prazosin is in the treatment of bulimic patients experiencing distressing nightmares using subjective and objective measures.

DETAILED DESCRIPTION:
To the investigators knowledge, there is no treatment trial for prazosin use in patients with bulimia nervosa struggling with nightmares, looking at either objective or subjective measures. The investigators plan to probe the effectiveness of prazosin in bulimic patients experiencing nightmares due to PTSD using both subjective and objective measures in order to improve future clinical care. The effects of prazosin on decreasing nightmares and bulimic symptoms on subjective scales and effects on sleep architecture using objective polysomnogram (PSG) measurements will help inform targeted psychopharmacologic and psychotherapeutic strategies to improve clinical care of bulimic patients struggling with distressing dreams secondary to PTSD. This study will be performed in two phases. Phase A will involve eight participants who will be tested using subjective scales (mentioned below). If Phase A data analysis leads to detection of a signal of efficacy 2 more participants will be recruited to participate in phase B of this trial using objective polysomnogram measurements. The results from this project will aid in establishing a fully powered clinical trial for treatment of nightmares in bulimic patients and improve outcomes in this high risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Clinical diagnosis of Bulimia Nervosa with complaint of nightmares secondary to PTSD

Exclusion Criteria:

* Restless leg syndrome
* Narcolepsy
* Sleep Apnea
* Neurological disorders
* Pregnancy
* cardiac abnormalities
* significant electrolyte abnormalities
* Use of steroids, beta blockers, prazosin
* Alcohol/substance abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07; Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fauzia Mahr, Principal Investigator — Penn State College of Medicine, Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Aurora RN, Zak RS, Auerbach SH, Casey KR, Chowdhuri S, Karippot A, Maganti RK, Ramar K, Kristo DA, Bista SR, Lamm CI, Morgenthaler TI; Standards of Practice Committee; American Academy of Sleep Medicine. Best practice guide for the treatment of nightmare disorder in adults. J Clin Sleep Med. 2010 Aug 15;6(4):389-401. PMID 20726290
- [Background] Singareddy R, Krishnamurthy VB, Vgontzas AN, Fernandez-Mendoza J, Calhoun SL, Shaffer ML, Bixler EO. Subjective and objective sleep and self-harm behaviors in young children: a general population study. Psychiatry Res. 2013 Oct 30;209(3):549-53. doi: 10.1016/j.psychres.2013.03.036. Epub 2013 Apr 23. PMID 23623452
- [Background] Dansky BS, Brewerton TD, Kilpatrick DG, O'Neil PM. The National Women's Study: relationship of victimization and posttraumatic stress disorder to bulimia nervosa. Int J Eat Disord. 1997 Apr;21(3):213-28. doi: 10.1002/(sici)1098-108x(199704)21:33.0.co;2-n. PMID 9097195
- [Background] Mitchell KS, Mazzeo SE, Schlesinger MR, Brewerton TD, Smith BN. Comorbidity of partial and subthreshold ptsd among men and women with eating disorders in the national comorbidity survey-replication study. Int J Eat Disord. 2012 Apr;45(3):307-15. doi: 10.1002/eat.20965. Epub 2011 Oct 19. PMID 22009722
- [Background] Gleaves DH, Eberenz KP, May MC. Scope and significance of posttraumatic symptomatology among women hospitalized for an eating disorder. Int J Eat Disord. 1998 Sep;24(2):147-56. doi: 10.1002/(sici)1098-108x(199809)24:23.0.co;2-e. PMID 9697013
- [Background] Bicanic IA, Postma RM, Sinnema G, De Roos C, Olff M, Van Wesel F, Van de Putte EM. Salivary cortisol and dehydroepiandrosterone sulfate in adolescent rape victims with post traumatic stress disorder. Psychoneuroendocrinology. 2013 Mar;38(3):408-15. doi: 10.1016/j.psyneuen.2012.06.015. Epub 2012 Aug 4. PMID 22867760
- [Background] Vgontzas AN, Tsigos C, Bixler EO, Stratakis CA, Zachman K, Kales A, Vela-Bueno A, Chrousos GP. Chronic insomnia and activity of the stress system: a preliminary study. J Psychosom Res. 1998 Jul;45(1):21-31. doi: 10.1016/s0022-3999(97)00302-4. PMID 9720852
- [Background] Lester NA, Keel PK, Lipson SF. Symptom fluctuation in bulimia nervosa: relation to menstrual-cycle phase and cortisol levels. Psychol Med. 2003 Jan;33(1):51-60. doi: 10.1017/s0033291702006815. PMID 12537036
- [Background] Ross RJ, Gresch PJ, Ball WA, Sanford LD, Morrison AR. REM sleep inhibition by desipramine: evidence for an alpha-1 adrenergic mechanism. Brain Res. 1995 Dec 1;701(1-2):129-34. doi: 10.1016/0006-8993(95)00984-x. PMID 8925274
- [Background] Taylor FB, Martin P, Thompson C, Williams J, Mellman TA, Gross C, Peskind ER, Raskind MA. Prazosin effects on objective sleep measures and clinical symptoms in civilian trauma posttraumatic stress disorder: a placebo-controlled study. Biol Psychiatry. 2008 Mar 15;63(6):629-32. doi: 10.1016/j.biopsych.2007.07.001. Epub 2007 Sep 14. PMID 17868655
- [Background] Germain A, Richardson R, Moul DE, Mammen O, Haas G, Forman SD, Rode N, Begley A, Nofzinger EA. Placebo-controlled comparison of prazosin and cognitive-behavioral treatments for sleep disturbances in US Military Veterans. J Psychosom Res. 2012 Feb;72(2):89-96. doi: 10.1016/j.jpsychores.2011.11.010. Epub 2011 Dec 20. PMID 22281448

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant consented to the study, but decided not to continue before completing screening measures due to scheduling difficulties.
Groups:
- Prazosin, Then Placebo: A starting dose of Prazosin (1mg capsule) will be given at Week # 1 of this arm. Symptoms will be reassessed and medication will be adjusted by 1-2 mg increments every 7 days for 3 weeks based on clinical response and severity of night mares, to achieve maximum therapeutic benefit while monitoring adverse effects using side effects scale on weekly basis (psychiatrist will be using the scale at every visit). The end point for capping the Prazosin dose will be 6 mg daily. After a washout period of 1 week, they then will receive matching placebo pill.
- Placebo, Then Pazosin: Placebo will be given for a 3 consecutive week period during the 7 week study period. After a washout period of 1 week, they then will be given Prazosin matched pill (1mg capsule). Symptoms will be reassessed and medication will be adjusted by 1-2 mg increments every 7 days for 3 weeks based on clinical response and severity of night mares, to achieve maximum therapeutic benefit while monitoring adverse effects using side effects scale on weekly basis (psychiatrist will be using the scale at every visit). The end point for capping the Prazosin dose will be 6 mg daily.
  Placebo: Placebo (sugar pill) is used for 3 weeks.
Period: First Intervention (3 Weeks)
Arm/Group | Prazosin, Then Placebo | Placebo, Then Pazosin
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Prazosin, Then Placebo | Placebo, Then Pazosin
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0
Period: Second Intervention (3 Weeks)
Arm/Group | Prazosin, Then Placebo | Placebo, Then Pazosin
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants received Prazosin (1mg capsule) and Placebo during the course of the research study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Weight (kg) [Mean (Standard Deviation); unit: Weight in (kg)] | 60.6 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Frequency of Nightmares Using the Sleep-50 Questionnaire
Description: The individual question about frightening dreams from the Nightmares Subscale of a self-administered questionnaire (Sleep-50 Questionnaire), will be used to determine if there is a decrease in frequency of nightmares in patients undergoing drug intervention. For each question, respondents are provided with a scale ranging from 1 ("not at all") to 4 ("very much") and are asked to indicate the extent to which the statement has matched their experience over the study time frame. The scale values range from 1-4, where a lower value indicates lower frequency of nightmares. A higher score is a worse outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Placebo will be given for a 3 consecutive week period during the 7 week study period.
  Placebo: Placebo (sugar pill) is used for 3 weeks.
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale | 2.25 (.37) | 2.75 (.25)

2. Primary Outcome: Decrease in Rapid Eye Movement (REM) Density & Normalization of REM Disruptions
Description: PSG (Polysomnogram) will be used in 2 participants to determine if there is a decrease in REM density in patients undergoing drug intervention.
Time Frame: 3 weeks
Population: This study was designed to include a second phase involving polysomnography in 2 participants if there was enough signal efficacy found based on subjective measures. The second phase was not done, therefore no data was analyzed for this outcome measure.
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Decrease in Bulimia Symptoms
Description: EDI-3 (Eating Disorder Inventory 3 Scale) is a pencil and paper test consisting of 91 items and 12 sub-scales. The main scales are the drive for thinness and the bulimia scales, the remaining sub-scales are: low self-esteem, body dissatisfaction, maturity fears, personal alienation, interpersonal alienation, interpersonal insecurity, perfectionism, interoceptive deficits, emotional dysregulation, and asceticism. The response options are based on a 6-point Likert-type scale are: Always, Usually, Often, Sometimes, Rarely, and Never. There are six composite scores, 12 primary scores, and three response style validity indicators. Software is used to calculate the raw scores, composite scores, validity scale scores and the T-scores. The t-score for the Bulimia scale will be used for this analysis with a range of 22-66. Higher scores indicate the likelihood of an eating disorder. A higher t-score on the bulimia scale indicates a worse outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: T-Score
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 8 | 8
T-Score | 43.1 (5.0) | 38.6 (4.8)

4. Secondary Outcome: Decrease in Total CAPS Score (PTSD)
Description: The CAPS (Clinician administered PTSD) rating scale consists of 30 questions rated on a 0-4 point scoring system and patient interview will be used to determine if there is a decrease in PTSD Symptoms among participants undergoing drug intervention. 17 of these questions are used to calculate the total severity score used in this analysis. This is done by summing the frequency and intensity ratings (each ranging from 0-4) for each of the 17 questions. The total severity score can have a range of 0-136. A higher score on this scale indicates a worse outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale | 65.5 (9.1) | 79.8 (12.9)

5. Secondary Outcome: Decrease in Depressed Mood as Measured by the HDRS (Hamilton Depression Rating Scale) and Subject Interview
Description: Rating scales and subject interview will be used to determine if there is a decrease in depressed mood among participants undergoing drug intervention. The HDRS (Hamilton Depression Rating Scale) consists of 17 items, some scored on a 5-point scale (0-4) and others scored on a 3-point scale (0-2). Items from the scale can be summed to give a total score ranging from 0 to 50, with higher scores indicating a worse outcome. This analysis is based on a single item from the scale (Depressed Mood, measured on a 5-point scale) where a higher score again indicates a worse outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale | 1.4 (0.4) | 1.3 (.50)

6. Secondary Outcome: Decrease in Self Harm Thoughts as Measured by the HDRS and Subject Interview
Description: Rating scales and subject interview will be used to determine if there is a decrease in self harm among participants undergoing drug intervention. The HDRS (Hamilton Depression Rating Scale) consists of 17 items, some scored on a 5-point scale (0-4) and others scored on a 3-point scale (0-2). Items from the scale can be summed to give a total score ranging from 0 to 50, with higher scores indicating a worse outcome. This analysis is based on a single item from the scale (Self Harm, measured on a 5-point scale) where a higher score again indicates a worse outcome.
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale | 0.5 (0.4) | .1 (.1)

ADVERSE EVENTS:
Time Frame: 2 years, 1 month.
Arm/Group | Prazosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT02382848/Prot_SAP_000.pdf